CLINICAL TRIAL: NCT04431349
Title: Comparison of Coronary Artery Bypass Graft Surgery Related Bleeding Complications in Patients Treated With Ticagrelor or Clopidogrel
Brief Title: Comparison of CABG Related Bleeding Complications in Patients Treated With Ticagrelor or Clopidogrel
Acronym: CABG
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, Assistant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-19-434
Record Dates: First submitted 2020-05-07; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Blood Loss, Surgical; Ticagrelor; Clopidogrel
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ticagrelor: The patient with acute myocardial infarction received loading dose of ticagrelor for coronary angiography within 2 days prior to OPCAB or CABG.
  Interventions: Drug: Ticagrelor 180mg
- clopidogrel: The patient with acute myocardial infarction received loading dose of clopidogrel for coronary angiography within 2 days prior to OPCAB or CABG.
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Ticagrelor 180mg — Patient received loading dose of ticagrelor for coronary angiography within 2 days prior to OPCAB or CABG.
  Groups: ticagrelor
Drug: Clopidogrel 75mg — Patient received loading dose of clopidogrel for coronary angiography within 2 days prior to OPCAB or CABG.
  Groups: clopidogrel

SUMMARY:
In patients with coronary artery disease, dual antiplatelet therapy (acetylsalicylic acid and a P2Y12-receptor antagonist) is a commonly used method because of its excellent antithrombotic effect. In particular, in patients with acute myocardial infarction, who receive coronary angiography as an emergency, the dual antiplatelet is used immediately before the test to prevent and test further clot formation, regardless of whether or not the patient had previously taken dual antiplatelet.

Ticagrelor, a direct-acting and reversible ADP receptor antagonist, was introduced in Denmark in 2013 and is now the most commonly used ADP receptor antagonist in the treatment of ACS. Compared to its predecessor clopidogrel, the pharmacokinetic proﬁl of ticagrelor is more predictable, demonstrating a faster onset of action and a more consistent platelet inhibition. However, because of the excellent antithrombotic effect and increased bleeding potential, it is recommended that major bleeding, such as OPCAB or CABG surgery, be expected with a high probability, and in case of fatal surgery, the drug should be discontinued for 5 days.

Most patients who receive emergency coronary heart surgery after undergoing coronary angiography as an emergency due to an acute myocardial infarction, it take approximately 24-48 hours to undergo surgery after examination. In fact, there have been reports of large-scale cross-country studies that do not increase bleeding risk compared to 5 days until 3 days after ticagrelor is stopped. Therefore, this study aimed to retrospectively analyze the bleeding tendency by analyzing the records of patients using clopidogrel or ticagrelor in preoperative coronary angiography for patients undergoing emergency CABG surgery from 2016 to September 2019.

ELIGIBILITY:
Inclusion Criteria:

* The patient with acute myocardial infarction received loading dose of clopidogrel or ticagrelor for coronary angiography within 2 days prior to emergency OPCAB or CABG.

Exclusion Criteria:

* heart surgery combined with other operation (valve surgery, aorta surgery, trauma surgery)
* History of coagulopathy
* History of liver cirrhosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency OPCAB or CABG surgery in Ajou university hospital from January 2016 to September 2019
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Major bleeding event | within 48hours after operation
  major bleeding defined as BARC-CABG related bleeding

SECONDARY OUTCOMES:
RBC transfusion amount | through study completion, an average of 1 month
  total amount of RBC transfusion within hospital stay after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No